CLINICAL TRIAL: NCT00682201
Title: Hemodynamic Changes During Normal Pregnancy: A Prospective Cohort Study of 100 Healthy Pregnant Women
Brief Title: Hemodynamic Changes During Normal Pregnancy
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Øyvind Skraastad, Head of The Division of Anaesthesia and Intensive Care Medicine, Rikshospitalet University Hospital, Oslo, Norway
Other Study IDs: storkhemo-08-GG
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-06

CONDITIONS: Pregnancy
Keywords: Pregnancy; Blood pressure; Cardiac output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Healthy pregnant women

SUMMARY:
Prospective, observational study of the changes in hemodynamic variables such as blood pressure, cardiac output, systemic vascular resistance, and of changes in respiratory variables such as vital capacity, and functional residual volume.A cohort study of 100 healthy pregnant women tested with non-invasive methods during pregnancy and 6 months after delivery.

DETAILED DESCRIPTION:
Healthy pregnant women with the willingness to consent in physiologic tests at 3 different time points during, and one time point after pregnancy. Spirometric tests will be performed with V-MAX, non-invasive measuring of hemodynamics will be measured by Finometer.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who at first admission are healthy

Exclusion Criteria:

* Co-existing diseases who represents decreased physical or psychological function

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healty pregnant women scheduled for delivery at the Birth Clinic, Rikshospitalet University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy specific changes in hemodynamic variables | Normal pregnancy time frame

SECONDARY OUTCOMES:
Respiratory functional changes | Normal pregnancy time frame

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, PhD MD, Study Director — Rikshospitalet University Hospital
Locations (1):
- Rikshospitalet University Hospital, Division of Anesthesia and Critical Care Medicine, Oslo, Norway